CLINICAL TRIAL: NCT04130399
Title: Study of Neoadjuvent Chemotherapy Followed by SBRT in Patients With Resectable and Borderline Resectable Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is being abandoned.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Susannah Ellsworth, Assistant Professor of Radiation Oncology, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0686
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cancer; Pancreatic Adenocarcinoma
Keywords: Folfirinox; Cancer; Radiation Therapy; neoadjuvent chemotherapy; Stereotactic Body Radiation Therapy (SBRT)
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Radiosurgery; folfirinox

STUDY DESIGN:
Intervention Model Description: preoperative chemotherapy with FOLFIRINOX followed by SBRT in patients with resectable pancreatic cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Preoperative Chemotherapy + SBRT (Experimental): Participants in this trial will receive neoadjuvant and adjuvant FOLFIRINOX chemotherapy for 6 cycles (1 cycle = 14 days) per routine guidelines.
  After 6 cycles of neoadjuvant therapy are completed, patients will undergo imaging with pancreatic protocol CT and PET-MRI to assess disease status . Patients without evidence of disease progression at the end of 6 cycles of neoadjuvant treatment will proceed to SBRT followed by surgical resection.
  Following surgery, patients will receive an additional 6 cycles of FOLFIRINOX chemotherapy.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: FOLFIRINOX

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Patients will receive 5 fractions of SBRT delivered over a five-day period. Treatment may be delivered over 2 weeks, provided that the patient receives at least 2 fractions per week.
Drug: FOLFIRINOX — Participants in this trial will receive neoadjuvant and adjuvant FOLFIRINOX chemotherapy for 6 cycles (1 cycle = 14 days) per routine guidelines

SUMMARY:
The purpose of this study is to research the effects of delivering full-dose neoadjuvant multi-agent chemotherapy (folfirinox) followed by stereotactic body radiation therapy (SBRT) in patients with resectable pancreatic ductal adenocarcinoma (PDAC) in order to intensify local therapy and improve outcomes.

DETAILED DESCRIPTION:
Primary Objectives:

1. To assess one-year local control rates in patients with operable PDAC who receive neoadjuvant chemotherapy and SBRT

Secondary Objectives:

1. To assess the following disease control endpoints: pathological response, disease-free survival, overall survival, failure pattern (local vs. distant) and time to development of distant metastases
2. To assess safety of the SBRT regimen

Exploratory objectives

1. To obtain exploratory data correlating tumor response grade with changes in circulating tumor DNA levels following chemotherapy, SBRT, and surgery in patients with PDAC
2. To obtain exploratory data correlating circulating tumor DNA (ctDNA) changes with disease control endpoints (overall survival, disease-free survival, failure pattern, and time to development of distant metastases)
3. To obtain exploratory data on positron emission tomography (PET) and magnetic resonance imaging (MRI) findings and correlations with tumor response among patients treated on study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Pathologic confirmation of pancreatic ductal adenocarcinoma
3. Resectable disease (determined by treating surgeon)
4. Patients planning to receive neoadjuvant Folfirinox as part of their standard of care treatment
5. No evidence of distant organ metastatic disease
6. Eastern Cooperative Oncology Group Performance status 0-1
7. Ability to understand and the willingness to sign informed consent document
8. Adequate organ function, defined by the following laboratory values, at the time of study entry:

   1. Hemoglobin ≥ 10 g/dL (transfusions acceptable)
   2. Absolute Neutrophil Count ≥ 0.5 x 109/L
   3. Platelets ≥ 100 x 109/L
   4. Creatinine ≤ 1.5x institutional upper limit of normal (ULN) or creatinine clearance ≥ 50 mL/min
   5. Total bilirubin ≤ 2x institutional ULN
   6. Aspartate aminotransferase test (AST)/ Alanine Aminotransferase Test (ALT) ≤ 3x institutional ULD

Exclusion Criteria:

1. Severe/uncontrolled intercurrent illness that, in the opinion of the patient's treating physicians, would prevent the patient from receiving either multi agent chemotherapy, high-dose radiation, or undergoing resection of the pancreatic tumor
2. Prior therapy for PDAC
3. Prior radiation to the upper abdomen (RT to other sites acceptable)
4. Inability to undergo port or PICC line placement
5. Active gastric or duodenal ulcer
6. Tumor invasion of the intestinal or gastric lumen
7. Active hepatitis B or other active serious infections
8. Pregnant and breastfeeding women are excluded. Women of child-bearing potential must have a negative urine or serum pregnancy test and be willing to use acceptable methods of birth control (hormonal or barrier method of birth control; abstinence) to avoid pregnancy for the duration of the study treatment
9. Life expectancy of < 3 months
10. Patients with contraindications to either PET scan or MRI (e.g., pacemaker/ICD) will NOT be excluded from study participation. Such patients will be treated per protocol but will not be required to undergo PET-MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Local control rate among PDAC patients treated with neoadjuvant chemotherapy followed by SBRT | 1 year after surgery date

SECONDARY OUTCOMES:
Pathological tumor response grade | Surgery Date (4 weeks [+/- 14 days] from end of SBRT)
Rate of margin negative resection | Surgery Date (4 weeks [+/- 14 days] from end of SBRT)
Rate of progression free survival | From surgery date to first documented date of progression, up to 5 years
Overall survival | From surgery date to date of death, up to 5 years
Local control rate | from date of surgery until date of first documented local failure, up to 5 years
Time to development of distant metastases | From surgery date to date of first documented metastatic disease, up to 5 years
Site of first failure | From surgery date to date of first documented metastatic disease, up to 5 years
Rate of grade 3-4 non hematological toxicity rates | Date of first fraction of SBRT through 30 days (+/-14) after surgery date

CONTACTS AND LOCATIONS:
Overall Officials: Susannah Ellsworth, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States